CLINICAL TRIAL: NCT06506695
Title: Optimizing Surgical and Prosthetic Workflow for Implant-supported Ear and Nose Prostheses With Early Loading and Distant Prosthesis Fabrication: A Prospective Cohort Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2024-0171
Record Dates: First submitted 2024-05-01; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Facial Deformity; Implant Complication
Keywords: Facial defect; Facial Prosthesis; Ear prosthesis; Nose prosthesis; Craniofacial implant; Anaplastology; Prosthesis fabrication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early loading of craniofacial prosthesis (Experimental)
  Interventions: Device: Craniofacial implant placement

INTERVENTIONS:
Device: Craniofacial implant placement — * Resection of oncologic process or remnants after trauma if necessary
  * Placement of craniofacial implants in the nasal floor and/or the temporal bone.
  * Placement of split thickness skin graft around the implants
  * Placement of nose and/or ear prosthesis within 3 weeks

SUMMARY:
Facial defects created by trauma, oncological procedures or congenital conditions can be repaired with ear, nose and/or eye prostheses. These are fixed on intraosseous implants placed in the temporal, nasal and orbital bone. To date, an osseointegration period of 3-6 months is maintained after which the implants are loaded.

This study aims to achieve two goals:

1. To load the implants with a nose or ear prosthesis within one month (preferably <3 weeks). Patients with an orbital prosthesis will not be recruited. In other words, an optimization of an existing protocol will be investigated. The quality of life of the patients as well as possible complications of the implants will be investigated.
2. Because of the short time between the surgery and the placement of the prosthesis, the prosthesis will be fabricated remotely. This means that the patient will not have to travel to the prosthetist. The feasibility and aesthetics will be analyzed through questionnaires for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a facial defect in the nasal and/or temporal area that will not be repaired with autologous tissue;
* Adult patients receiving oncological resection or trauma resulting in a facial defect in the nose and/or ear that will not be repaired with autologous tissue;
* Patients who can come to the hospital every week for 6 weeks.

Exclusion Criteria:

* Patients with insufficient bone mass for implant placement
* Patients who cannot come to the hospital for weekly follow-ups
* Patients that wish an autologous reconstruction
* Patient is unable to tolerate general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of implant survival in nasal and temporal bone from 0-100% | 6 months after placement of implants
  Investigate craniofacial implant survival. 100% being better than 0%.
Peri-implant complications using the Holgers' (grade 0-4) | 6 months after placement of implants
  Investigate craniofacial peri-implant complications after early loading concept using the Holgers' scale from 0, meaning excellent peri-implant status to 4 necessitating removal of the implant.
Peri-implant complications using the IPS scale (IPS-score) | 6 months after placement of implants
  Investigate craniofacial peri-implant complications after early loading concept using the IPS scale. Only the 'percutaneous' part of the scale will be used. IPS scale ranges from no treatment to removal of the implant.
Quality of Life with SF-36, SWLS and RSES and self-made questionnaire | Before treatment and 6 months after implant placement
  Assessing the patient's quality of life using the early loading protocol with standardised and self-made questionnaires. The SF-36 scoring will result in 8 scales ranging from 0-100 with the lower the score the more disability. SWLS will result in a range of 5-35. The higher the score the higher the satisfaction with life. RSES ranges from 0-30. Scores between 15 and 25 are considered in the normal range whereas scores below 15 suggest low self-esteem. The self-made questionnaires will result in percentages of the given answers.

SECONDARY OUTCOMES:
Difference in surface matching of the midface and temporal area in mm | 6 months after implant placement
  By matching and comparing surface scans we can analyse the swelling in the midface and temporal area after directly after surgery and postoperatively. These will result in positive or negative changes and expressed in millimeters.
Implant stability over time with implant stability quotient (ISQ) range 1-100 | 6 months after implant placement
  By measuring stability we can create an osseointegration timeline for craniofacial implants. Higher values indicate higher stability. Values in between 55 and 85 are considered acceptable.
Feasibility of remote prosthesis fabrication | 6 months after implant placement
  Questionnaires assessing the experience of the patient and aesthetics of the prosthesis

IPD SHARING:
Plan to Share IPD: Yes
Anonymized raw data will be shared with the scientific community. All materials that can be used to identify the patient such as face scans and clinical pictures will not be shared.
Supporting Information: Study Protocol, CSR
Time Frame: After study publication for a time period of 5 years
Access Criteria: Data can be requested via mail to the PI: matthias.ureel@uzgent.be